CLINICAL TRIAL: NCT05983666
Title: POCUS ASSESSMENT FOR TRACHEAL VS OESOPHAGEAL INTUBATION
Acronym: PATO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Clinica Universidad de Navarra, Universidad de Navarra (Other)
Responsible Party: Sponsor
Other Study IDs: PATO
Record Dates: First submitted 2023-07-24; First posted 2023-08-09 (Actual); Last update posted 2023-08-09 (Actual); Status verified 2023-06

CONDITIONS: Intubation Complication
Keywords: Tracheal intubation; Ultrasound

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients undergoing scheduled and/or emergency surgery requiring orotracheal intubation.
  Interventions: Diagnostic Test: Ultrasound Oesophageal Intubation

INTERVENTIONS:
Diagnostic Test: Ultrasound Oesophageal Intubation — Ultrasound Oesophageal intubation detection

SUMMARY:
The clinical importance of airway management has gained prominence in the last decade in most scientific societies with the aim of improving the standard of care.

The WHO has focused guidelines for "Safety in Surgery", which attempt to encompass all methods that predict and recognise airway management risk and should be applied by the surgical team, and has therefore created and implemented a surgical checklist that can be useful in reducing the risk of unidentified difficulties.

The same suggestion has been included in the Helsinki Declaration on Patient Safety in Anaesthesiology, signed by most European entities in cooperation with the European Society of Anaesthesiology (ESA), the European Board of Anaesthesiology (EBA-UEMS), and the World Federation of Societies of Anaesthesiology (WFA).

Confirmation of correct endotracheal tube (ET) placement is a crucial step in airway management, as unrecognised oesophageal intubation can have catastrophic consequences. Numerous methods are used to verify correct ET placement, including visual confirmation of tube passage through the vocal cords during laryngoscopy, chest wall expansion during ventilation, visualisation of the tracheal rings and carina using a flexible bronchoscope, auscultation, capnometry, capnography and chest radiography. These techniques vary in their degree of precision. Although capnography is considered the gold standard for confirming tracheal intubation, it has some important limitations.

In recent years, ultrasonography has been introduced as the fifth pillar of the physical examination of the patient: inspection, palpation, percussion, auscultation and insonation. For airway assessment and management, Point-of-Care UltraSound (PoCUS) has been incorporated into routine clinical practice, answering open diagnostic questions, aiding in differential diagnosis and guiding procedures.

Thus, investigators propose a simple, quick and easy-to-learn approach for the interpretation of ultrasound imaging findings during airway management.

DETAILED DESCRIPTION:
The first step of the algorithm is to locate the oesophagus by asking the patient to swallow. The ultrasound transducer is placed transversely on the anterior surface of the neck at the paratracheal level (usually located on the left side), 1-2 cm above the sternal notch or jugulum. In this image, the trachea is shown as a hyperechoic, curvilinear image (air-mucosa interface), showing a posterior reverberation artefact called a comet tail. During the intubation technique, this ultrasound window allows the physician to observe the real-time passage of the tube into the trachea, confirming correct tracheal intubation only if a single air-mucosa interface with its comet tail is maintained. This can then be verified by capnography (if available) or by lung sliding.

ELIGIBILITY:
Inclusion Criteria:

Patients (male or female) ASA I-III, aged between 18 and 90 years, undergoing scheduled and/or emergency surgery requiring orotracheal intubation. Informed consent form must be signed authorising inclusion in the study.

Exclusion Criteria:

A.- Cervical tumours, goitre or patients who have required cervical radiotherapy.

B.- Abnormalities leading to alterations of the anatomy such as facial/cervical fractures.

C.- Those who cannot give their consent.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients (male or female) ASA I-III, aged between 18 and 90 years, undergoing scheduled and/or emergency surgery requiring orotracheal intubation. Informed consent form must be signed authorising inclusion in the study.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-07-01 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
Ultrasound Oesophageal Intubation | 5 minutes
  To assess a diagnostic algorithm for tracheal versus oesophageal intubation using ultrasound and capnography as a confirmatory criterion.

SECONDARY OUTCOMES:
POCUS learning curve | 30 minutes
  Time required for the application of the ultrasound algorithm and training time for previously untrained personnel.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinica Universidad de Navarra, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No
It is not neccessary to share any data.